CLINICAL TRIAL: NCT00392860
Title: Development of an Ergonomic Manual Wheelchair Pushrim- Phase II
Brief Title: Development of an Ergonomic Wheelchair Pushrim
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michael Boninger, Chair, Department of Physical Medicine and Rehabilitation, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02484, 0511136
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-01

CONDITIONS: Spinal Cord Injury
Keywords: Wheelchair; Handrims; Rehabilitation; Upper extremity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- PalmRim Experimental (Experimental): Participants will have PalmRim installed on their wheelchair.
  Interventions: Device: PalmRim
- Natural-Fix Experiment (Experimental): Participants will have a Natural-Fit installed on their wheelchair.
  Interventions: Device: Natural-Fit
- Handrim Control (Placebo Comparator): Participants in this arm had a new standard handrim installed on their wheelchair as a control.
  Interventions: Device: Handrim Control Group

INTERVENTIONS:
Device: Natural-Fit — Ergonomic handrim for wheelchairs
  Arms: Natural-Fix Experiment
Device: PalmRim — Ergonomic handrim for wheelchair
  Arms: PalmRim Experimental
Device: Handrim Control Group — Participants were given a new standard handrim to test. This intervention group is the control group.
  Arms: Handrim Control

SUMMARY:
The purpose of this study is to test the effectiveness of newly designed ergonomic manual wheelchair handrims called the Natural-Fit and PalmRim when compared to a new standard handrim. It is our hope that the new design of the handrims will help reduce upper extremity pain and injury, which is very common among manual wheelchair users. The Natural-Fit handrim was designed to directly address the shortcomings of standard handrims and to improve the standard-round tube handrims which were designed over 50 years ago. The PalmRim was designed for individuals who have limited hand function, making it difficult to grasp standard handrims.

DETAILED DESCRIPTION:
This research will have three parts.

The first part will include completing propulsion and braking tasks with the subject's original handrims. After the initial testing, new handrims (NaturalFit, PalmRim, and a new standard handrim) will be installed on the subject's wheelchair and subjects will again be asked to complete another set of propulsion and braking tasks. Subjects will also be asked to complete a questionnaire to assess wrist and shoulder pain and undergo an examination of the condition of the palm of their hand.

For the second part of the study, subjects will be asked to participate in a 4-month trial use period of the new handrims on their wheelchair.

In the third part of the study, subjects will complete the final set of propulsion and braking tasks and complete a follow-up questionnaire.

ELIGIBILITY:
Natural-Fit

Inclusion Criteria:

* Use of a manual wheelchair as a primary means of mobility (over 40 hours per week)
* Use a standard handrim
* Between the ages of 18 and 55
* Has normal hand function

Exclusion Criteria:

* Pressure Sores

PalmRim

Inclusion Criteria:

* Use of a manual wheelchair as a primary means of mobility (over 40 hours per week)
* Use a vinyl-coated handrim
* Between ages 18 and 55
* Has impaired hand function

Exclusion Criteria:

* Pressure sores

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Boninger, MD, Principal Investigator — University of Pittsburgh and VA Pittsburgh Healthcare System
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from November 7, 2008 to April 8, 2009.
Pre-assignment Details: The manufacturer of the PalmRim decided not to pursue the design and development of the product. As a result, the PalmRim experiment arm did not enroll any participants.
Groups:
- Natural-Fit Experiment: Participants will have a Natural-Fit handrim installed on their wheelchair. The Natural-Fit device was designed to directly address the shortcomings of standard handrims and to improve the standard round-tube handrims which were designed over 50 years ago.
  Participants used the Natural-Fit Handrim for a four month trial period, before returning for follow up evaluations.
  Natural-Fit : Ergonomic handrim for wheelchairs
- PalmRim Experiment: Participants will have a PalmRim handrim installed on their wheelchair. The PalmRim was designed for individuals who have limited hand function, making it difficult to grasp standard handrims.
  Participants were to use the PalmRim handrim for a four month trial period, before returning for follow up evaluations.
- Handrim Control Group: Participants will be given a new standard handrim.
Period: Overall Study
Arm/Group | Natural-Fit Experiment | PalmRim Experiment | Handrim Control Group
Started | 3 | 0 | 1
Completed | 3 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Natural-Fit Experiment: Participants will have a Natural-Fit installed on their wheelchair.
  Natural-Fit : Ergonomic handrim for wheelchairs
- Control Group: Participants will be given a new standard handrim.
- Total: Total of all reporting groups
Arm/Group | Natural-Fit Experiment | Control Group | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (2.11) | 39 (0) | 46 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Status Score
Description: The Functional Status Scale, which measures hand and wrist symptoms.
Time Frame: Baseline, 4 Months
Population: Zero participants were analyzed because only 4 participants were enrolled in this trial. Analyzing the results would not result in any meaningful information. The manufacturer of the PalmRim decided not to pursue the design and development of the product. As a result, the PalmRim experiment arm did not enroll any participants.
Groups:
- Natural-Fit Experiment: Participants will have a Natural-Fit handrim installed on their wheelchair.
  Natural-Fit : Ergonomic handrim for wheelchairs
Arm/Group | Natural-Fit Experiment | Handrim Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Natural-Fit Experiment | Control Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No